CLINICAL TRIAL: NCT06000202
Title: Elastographic Improvement of Vaginal Atrophy Treated by Er:YAG Laser
Brief Title: Elastographic Improvement of Vaginal Atrophy Treated by Erbium Yag Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Cemal Tamer Erel, Prof. Principal investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 689852
Record Dates: First submitted 2023-08-12; First posted 2023-08-21 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Vaginal Atrophy; Dyspareunia; Laser; Genitourinary Syndrome of Menopause (GSM)
MeSH Terms: conditions — Dyspareunia

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participant doesn't know if she receives the sham or laser therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser Arm (Experimental): Non-ablative thermal-only Er:YAG laser (Fotona Dynamis) treatment using R11 and PS03 handpieces
  Interventions: Device: Fotona Dynamis Er:YAG Laser System
- Sham Arm (Sham Comparator): The same procedure is applied but with a sham handpiece.
  Interventions: Device: Sham

INTERVENTIONS:
Device: Fotona Dynamis Er:YAG Laser System — The patient receives 2940 nm Er:YAG Laser (XS Dynamis, Fotona, Slovenia) at intervals of 21 days. She receives 3 sessions, in total. Each session consists of application of PS03 handpiece intravaginal with spot size of 7 mm, fluence of 10 j/cm2, frequency of 1.6 Hz and 4-7 pulses per point and 6 passes followed by R11 handpiece intravaginal with spot size of 7 mm, fluence of 10 j/cm2, frequency of 1.6 Hz and 4-7 pulses per point and 3 passes.
  Arms: Laser Arm
Device: Sham — Er:YAG laser is applied with sham handpiece.
  Other Names: Placebo
  Arms: Sham Arm

SUMMARY:
This study is a randomized controlled sham applied study. Its aim is to evaluate the efficacy of Er:YAG laser for the treatment of atrophic vaginitis in postmenopausal women.

In this study, demonstration of the efficacy of Er:YAG laser for the treatment of atrophic vaginitis in postmenopausal women is intended with Maturation Index (MI), vaginal pH measurement, Female Sexual Function Index (FSFI), Vaginal Health Index (VaHI), Visual Analogue Scale (VAS) and ultrasonographic elastography

DETAILED DESCRIPTION:
In the postmenopausal period, especially due to estrogen deficiency, vaginal atrophy occurs in the vulvo-vagina, lower urinary tract, pelvic floor muscles and endopelvic fascia. Vaginal dryness secondary to atrophy in genital organs, pain and tenderness especially during sexual intercourse, and decreased genital elasticity are the most common symptoms and signs during the postmenopausal period. With regard to the urinary system, frequent urination, feeling of urgency, recurrent urinary tract infections, organ prolapses-urethrocele, cystocele, urethral prolapse and stress or urge type urinary incontinence could be seen.These signs and symptoms were recognized in 2014 by the International Society for the Study of Women's Sexual Health (ISSWSH) and the North American Menopause Society (NAMS) under the main title OF "genito-urinary syndrome of menopause" (GSM). During the postmenopausal period, a detailed history should be taken, a complete physical examination should be performed, and various tests should be performed for the evaluation of GSM.

Laser is a treatment option for the genitourinary symptoms that could occur at the postmenopausal period. Laser can be applied to vulva by giving an external beam, or it can be applied intravaginally or directly to the urethra using vaginal and urethral cannula.

The smooth mode application of the Er:YAG laser ensures that the laser beam retains the heat it gives without ablation and penetrates deeper into the tissue. After laser application, thermomechanical and thermochemical effects occur in the tissue, respectively. It provides controlled thermal energy and causes shrinkage of the collagen fibrils in the vaginal epithelium and lamina propria. It also induces neocollagenesis, elastogenesis and neoangiogenesis by temperature change. With minimum damage to the peripheral tissue, the viable cells in the target tissue reacts to this temperature change by expressing heat shock proteins (HSP). Then, HSP increases the levels of transforming growth factor-beta, fibroblast growth factor, epidermal growth factor, platelet-derived growth factor, vascular epithelial growth factor which induce neocollagenesis and neoangiogenesis. Therefore, the thermal energy stored in the vaginal wall induces proliferation of the epithelium which is rich in glycogen, neovascularization and collagen production in the lamina propria.

In this study, evaluation and demonstration of the efficacy of Er:YAG laser for the treatment of atrophic vaginitis in postmenopausal women is intended with Maturation Index (MI), vaginal pH measurement, Female Sexual Function Index (FSFI), Vaginal Health Index (VaHI), Visual Analogue Scale (VAS) and ultrasonographic elastography.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with vaginal atrophy symptoms
* Adult Female, 18 years of age or older

Exclusion Criteria:

* Patients with a history of previous vaginal operation,
* Patients with pelvic organ prolapse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 18 years and older postmenopausal women
Enrollment: 20 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Efficacy: Rate of improvement in vaginal atrophy | 6 months
  Evaluation of the efficacy and safety of vaginal atrophy by using ultrasonographic Elastography
Efficacy:Rate of improvement in sexual function | 6 months
  Evaluation of dyspareunia by Female Sexual Function Index
Efficacy: Rate of improvement in vaginal atrophy | 6 months
  Evaluation of Maturation Index
Efficacy: Rate of improvement in vaginal atrophy | 6 months
  Evaluation of Vaginal Health Index
Efficacy: Rate of improvement in pain | 6 months
  Evaluated by Visual Analogue Scale

SECONDARY OUTCOMES:
Safety:Incidence and severity of device related Adverse Events | 6 months
  Incidence and severity of device related Adverse Events (i.e., infections, edema, superficial burns, wound dehiscence)

CONTACTS AND LOCATIONS:
Overall Officials: Cemal Tamer Erel, Prof., Study Director — Istanbul University - Cerrahpasa
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul University-Cerrahpaşa, Istanbul
  - Istanbul University-Cerrahpasa, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
The results will be available after the completion of the study for a year.
Supporting Information: CSR
Time Frame: It will be available after the completion of the study for a year.

REFERENCES:
- [Derived] Bayraktar E, Erel CT, Akturk H, Erkan IBO, Hamid R, Alper E, Adaletli I, Urfalioglu M. A novel objective evaluation method, shear wave elastography, in the treatment of atrophic vaginitis by nonablative intravaginal Er:YAG laser, a randomized-sham controlled pilot study. Menopause. 2024 Aug 1;31(8):716-723. doi: 10.1097/GME.0000000000002380. Epub 2024 Jun 11. PMID 38860935